CLINICAL TRIAL: NCT03918161
Title: Magnetic Resonance Elastography of Transplanted Kidney (GREFFE_ELASTO IRM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2019/17
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Interstitial Fibrosis/Tubular Atrophy of Transplanted Kidneys
Keywords: Interstitial fibrosis; Tubular atrophy Renal transplantation; Renal allograft; Magnetic Resonance Imaging; Elastography; non-invasive diagnosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: All patients will realize Magnetic Resonance Elastography exam
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRE exam (Experimental): Magnetic Resonance Elastography (MRE) exam associated with standard T1-weighted and T2-weighted sequences
  Interventions: Device: MRE exam

INTERVENTIONS:
Device: MRE exam — Magnetic Resonance Elastography

SUMMARY:
: GREFFE_ELASTO IRM will evaluate Magnetic Resonance Elastography (MRE) in renal transplant patients with suspected interstitial fibrosis/tubular atrophy lesions requiring biopsy graft sampling under ultrasound control.

The main objective is to search a correlation between renal graft parenchymal elasticity values obtained in vivo by MRE, and the histological data of renal fibrosis by biopsy sampling, and providing a non-invasive tool capable of detecting and monitoring this development over time, making possible in the future to reduce the number of renal biopsies.

DETAILED DESCRIPTION:
The natural history of interstitial fibrosis/tubular atrophy (IF/TA) is a common mechanism of disease progression of transplanted kidneys. The process has been well studied through protocol biopsies. The early phase is characterized by fibrogenesis and the emergence of tubulo-interstitial damage due to immunologic phenomena; the late phase is characterized by the worsening of parenchymal lesions and the occurrence of glomerular sclerosis leading to graft loss.

Today, non-invasive markers of these pathological changes are missing and the protocol biopsies are still the only reliable tool for the diagnosis of IF/TA.

Elasticity imaging has already been proven in the management of chronic liver diseases with Fibroscan. In the field of renal diseases, several studies have been carried out in ultrasound elastography on renal grafts but the renal elastography is more difficult due to the complexity of the kidney (deep organ, two compartments, high vascularity). All these parameters have an influence on the elasticity measures.

The elastography imaging is also performed in MRI (Magnetic resonance imaging): The Magnetic Resonance Elastography (MRE). MRE is less subject to variations in depth, to the experience of the operator and to allow an overall evaluation of the graft.

The potentially eligible patients will be recruited by the nephrologist during a consultation in which renal biopsy is scheduled (as part of current practice). Patients meeting the inclusion criteria and having no exclusion criteria will be offered to participate in this study. If accepted, the only examination specific to this research, the MRE, will be scheduled to be performed the same day as the renal biopsy.

This MRE is painless, non-irradiating, and does not require the injection of contrast medium.

The participation of the patient ends when he leaves the hospital after the biopsy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18yrs;
* Transplanted kidney patient with suspicion of IF/TA lesions requiring biopsy graft sampling under ultrasound control;
* Signed informed consent;
* Affiliated or beneficiary of health insurance

Exclusion Criteria:

* Patients with dilated pyelocaliceal cavities on ultrasound or significant renal artery stenosis (> 80%) on Doppler;
* Pregnant or nursing women;
* Contraindications to MRI;
* Person deprived of liberty, major who is the subject of a legal protection measure or unable to express consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Mean value of renal elasticity | Baseline (defined as during MRE exam)
  5 times' measures in comparison with the upper pole of the graft which corresponds to the biopsy site (unit kilo-Pascal)

SECONDARY OUTCOMES:
Average value of renal elasticity | Baseline (defined as during MRE exam)
  measured in 10 areas of the graft Intra-renal inflammation, tubulitis, chronic vascular and glomerular lesions measured semi-quantitatively by the pathologist following the Banff classification

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No